CLINICAL TRIAL: NCT04749706
Title: Management of Constitutional Thinness Through an Adapted Physical Activity Program, Whether or Not Associated With Food Supplementation. Interventional Study Compared to Matched Controls: NUTRILEAN + Study
Acronym: NUTRILEAN +
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2020 DUCLOS; 2020-A02565-34 (Other: 2020-A02565-34)
Record Dates: First submitted 2021-02-04; First posted 2021-02-11 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Healthy Normal Weight Women; Constitutionally Lean Women
Keywords: energy metabolism; body composition; physical training; constitutional leanness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal weight (Active Comparator): the normal weight women will receive the 12-week physical activity intervention and serve as a control group.
  Interventions: Behavioral: Physical training alone
- constitutionally lean women - Physical training only (Experimental): women will receive the 12-week physical activity intervention
  Interventions: Behavioral: Physical training alone
- constitutionally lean women - Physical training + proteins (Experimental): women will receive the 12-week physical activity intervention in addition to a protein supplementation
  Interventions: Behavioral: physical training + protein intake

INTERVENTIONS:
Behavioral: Physical training alone — The physical activity intervention will consist in 12 weeks of training composed of 3 sessions per week. The three sessions will be mainly composed of resistance training aiming at increasing body weight through increased fat free mass. The main muscle groups (lower limbs, upper limbs and trunk) will be trained. The intervention will be performed under the supervision of a specialized coach.
  Arms: Normal weight; constitutionally lean women - Physical training only
Behavioral: physical training + protein intake — The physical activity intervention will consist in 12 weeks of training composed of 3 sessions per week. The three sessions will be mainly composed of resistance training aiming at increasing body weight through increased fat free mass. The main muscle groups (lower limbs, upper limbs and trunk) will be trained. The intervention will be performed under the supervision of a specialized coach.
  15 women with constitutional leanness will, on top of the physical training, received a daily protein supplementation corresponding to 20 grams of proteins + 10 grams of Maltodextrine
  Arms: constitutionally lean women - Physical training + proteins

SUMMARY:
The main aim of the present study is to compare the effect of a 12-week physical activity program on body weight gain and body composition changes between normal weight and constitutionally lean individuals. The second objective will be to question the potential additional effect of a protein supplementation coupled to the physical training intervention on body wright and body composition in constitutionally lean women.

DETAILED DESCRIPTION:
After a medical inclusion visit, the participants will realize a maximal aerobic test at the university hospital as well as a body composition analysis, a blood sample will be taken, their resting metabolic rate will be assessed as well as their energy metabolism during a rectangular cycling exercise. Their muscle strength and architecture will be assessed. Their energy intake and eating habits will also be assessed as well as their diet-induced thermogenesis in response to a fixed and an ad libitum meal. Their sleep metabolism will also be assessed using the Dreem technology. Questionnaires will be used to evaluate their daily free living energy intake and accelerometers used to assess their daily physical activity level.

The participants will then perform a 12-week physical activity intervention with 15 of the 30 constitutionally lean one receiving a protein supplementation (randomly assigned). All the measures will be replicated at the end of the intervention as well as 6 weeks after

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria common to both groups

* Adult women aged 18 to 35, having a stable weight for at least 3 months.
* Body mass index (BMI) ≤ 17.5 kg / m2 (for the "constitutional thinness" group) or 20 kg / m2 ≤ BMI ≤ 25 kg / m2 (for the normal-weighted control group)
* Able to give informed consent to participate in research.
* Affiliation to a Social Security scheme.

Inclusion criteria specific to women with constitutional thinness

* BMI ≤ 17.5 kg / m2
* Weight stable for at least 3 months
* No eating disorder
* No biological markers of undernutrition
* Absence of secondary amenorrhea

Inclusion criteria specific to normo-weighted subjects

* 20 kg / m2 ≤ BMI ≤ 25 kg / m2
* Weight stable for at least 3 months
* No eating disorder
* No biological markers of undernutrition
* Absence of secondary amenorrhea

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Severe progressive disease
* Medical or surgical history judged by the investigator to be incompatible with this study
* Diabetes or any other pathology limiting the application of one or the other trial strategy
* History of cardiovascular and / or neuro-vascular pathology, and / or cardiovascular and / or neuro-vascular risk factors (excluding obesity / overweight)
* Surgical intervention in the previous 3 months
* Taking medications that may interfere with the results of the study
* Regular practice of intense physical activity (more than 3 physical activity sessions per week)
* Regular consumption of tobacco or alcohol
* Special diet
* Abnormal plasma levels of IGF-1, estradiol, free T3, cortisol and leptin (only for the "constitutional thinness" group)
* Persons under guardianship or subjects deprived of their liberty by judicial or administrative decision
* Person in a period of exclusion from another study
* Refusal of participation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12-11 (Estimated)

PRIMARY OUTCOMES:
Change in body weight from baseline | day 1, day 90, day 145
  body weight using a classical scale at different time : baseline, after the 12-week intervention and after 6 weeks of follow-up .
Change in fat mass composition | day 1, day 90, day 145
  fat mass will be assessed using DXA
Change in fat free mass composition | day 1, day 90, day 145
  fat free mass will be assessed using DXA

SECONDARY OUTCOMES:
Change in bone structure | day 1, day 90, day 145
  the bone structure will be assessed thanks to DXA and pQCT
Change in muscle strength | day 1, day 90, day 145
  muscle strength assessed thanks to isometric contraction using Biodex.
Change in muscle structure | day 1, day 90, day 145
  muscle structure assessed thanks to muscle echography
Change in aerobic capacities . | day 1, day 90, day 145
  aerobic capacities assessed using indirect calorimetry during a graded cycling exercise
Change in resting metabolic rate | day 1, day 90, day 145
  resting metabolic rate assessed using indirect calorimetry during 30 minute rest in a comfortable inclined chair. The is the energy expended at rest in Kilo-Joules.
Change in Insulin | day 1, day 90, day 145
  Insulin will be evaluated in blood sample
Change in glycaemia, . | day 1, day 90, day 145
  glycaemia will be evaluated in blood sample
Change in triglycerides | day 1, day 90, day 145
  triglycerides will be evaluated in blood sample
Change in cholesterol | day 1, day 90, day 145
  cholesterol will be evaluated in blood sample
Change in leptin | day 1, day 90, day 145
  leptin will be evaluated in blood sample
Change in ghrelin | day 1, day 90, day 145
  ghrelin will be evaluated in blood sample
Change in adiponectin | day 1, day 90, day 145
  adiponectin will be evaluated in blood sample
Change in thyroid hormones | day 1, day 90, day 145
  thyroid hormones will be evaluated in blood sample
Change in LipoxMax | day 1, day 90, day 145
  the point of maximal use of lipids during exercise will be assessed during a graded exercise composed of 4 stages of 6 minutes each, using indirect calorimetry.
Change in Energy intake | day 1, day 90, day 145
  Energy Intake will be assessed using a Three-day dietary report (self-reported)
Change in physical activity level measured with an accelerometer | day 1, day 90, day 145
  The time spent at low-moderate and vigorous physical activity will be assessed using a 7-day accelerometry record
Change in sleep metabolism assessed with the dreem technology captors | day 1, day 90, day 145
  sleep metabolism assessed during a complete night, using the Dreem technology captors that consists in a simple band around the head during the night.

CONTACTS AND LOCATIONS:
Overall Officials: Martine DUCLOS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France